CLINICAL TRIAL: NCT04991974
Title: Opioid Use Disorder Treatment Linkage at Sexual Health Clinics Using Buprenorphine
Acronym: OUTLAST-B
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Baltimore City Health Department (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01DA045724 (NIH); R01DA045724 (NIH)
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Patient Navigation; Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual Care (UC) (No Intervention): The UC Arm will include standard services from the sexual health clinic / city health department [at the time of the study, no standardized intervention for opioid use disorder treatment linkage].
- Patient Navigation (PN) (Active Comparator): The PN Arm will include all UC Arm services, with the addition of a Patient Navigator who will assist the participant in selecting a community OUD treatment program, facilitate an intake appointment, help to resolve barriers and coordinate OUD treatment entry, and support early retention in OUD treatment.
  Interventions: Behavioral: Patient Navigation
- Patient Navigation + Buprenorphine Initiation (PN+BUP) (Experimental): The PN+BUP Arm will include all PN Arm services, with the addition of meeting with the sexual health clinic's buprenorphine-waivered provider (typically a nurse practitioner) to initiate buprenorphine treatment, as a bridge until successful transfer to OUD treatment in the community. The standard buprenorphine bridge prescription will be for buprenorphine/naloxone film: 8/2mg, up to 16mg per day, 7 day supply.
  Interventions: Behavioral: Patient Navigation; Drug: Buprenorphine

INTERVENTIONS:
Behavioral: Patient Navigation — A Patient Navigator will work with participants to facilitate their entry into OUD treatment in the community (e.g., by selecting a program, scheduling intake appointments, and addressing barriers to facilitate successful treatment linkage).
  Arms: Patient Navigation (PN); Patient Navigation + Buprenorphine Initiation (PN+BUP)
Drug: Buprenorphine — Buprenorphine is an FDA-approved medication for opioid dependence, and will be used in this study consistent with its approved use (but will be initiated in the novel setting of sexual health clinics in this health services study).
  Participants will meet with an sexual health clinic provider who holds a waiver to prescribe buprenorphine. Participants will initiate buprenorphine treatment via a home induction under the direction of the provider. Because barriers to transfer may take some time to overcome, participants will be able to receive additional bridge buprenorphine up to two times (up to 15 days' supply at a time) until successful transfer to OUD treatment in the community.
  Other Names: Buprenorphine/naloxone sublingual film
  Arms: Patient Navigation + Buprenorphine Initiation (PN+BUP)

SUMMARY:
This study will examine the effectiveness of opioid use disorder (OUD) treatment linkage strategies for patients seen at sexual health clinics. This 3-arm RCT will compare Usual Care vs. Patient Navigation vs. Patient Navigation + Buprenorphine Initiation (UC vs. PN vs. PN+BUP).

DETAILED DESCRIPTION:
This study, entitled Opioid Use Disorder Treatment Linkage at Sexual Health Clinics using Buprenorphine (OUTLAST-B), will examine opioid use disorder (OUD) treatment linkage strategies for people receiving sexual health services from public clinics and health departments. This three-arm, parallel randomized clinical trial (RCT) will compare Usual Care (UC), vs. referral via Patient Navigation (PN), vs. Patient Navigation with buprenorphine initiation (PN+BUP).

The UC Arm will include standard services at the sexual health clinic / city health department.

The PN Arm will include all UC Arm services, with the addition of a Patient Navigator who will assist the participant in selecting a community OUD treatment program, facilitate an intake appointment, help to resolve barriers and coordinate OUD treatment entry, and support early retention in OUD treatment.

The PN+BUP Arm will include all PN Arm services, with the addition of meeting with the sexual health clinic's buprenorphine-waivered provider (typically a nurse practitioner) to initiate buprenorphine treatment, as a bridge until successful transfer to OUD treatment in the community.

Research assessments consisting of a structured interview battery and biomarkers for drug use and sexually transmitted infections will be conducted at baseline, 3-, and 6-month follow-up. Selected outcomes will be examined through 12-months via health record linkage methods. The study will examine participant outcomes in the domains of: (1) OUD treatment entry and retention, (2) Opioid use and related problems (including fatal and non-fatal overdose), and (3) HIV/STD-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Opioid use in the past 30 days
3. DSM-5 diagnostic criteria for OUD with physiological dependence
4. Willing to try buprenorphine treatment.

Exclusion Criteria:

1. current enrollment in OUD treatment with buprenorphine, methadone, or extended-release naltrexone
2. clinical contraindication with buprenorphine (e.g., allergy to buprenorphine or naloxone, chronic pain management with opioid agonists)
3. regular use of illicit long-acting opioid agonists (e.g., methadone; due to potential challenges with dose induction)
4. heavy alcohol use that, in the judgement of the prescribing provider, raises a safety concern that precludes eligibility for buprenorphine induction
5. high dose or intravenous benzodiazepine misuse
6. pregnancy (due to special needs; will be treated outside of the study)
7. unstable medical or psychiatric illness (e.g., psychosis or active suicidal ideation)
8. inability to provide informed consent (e.g., failure to pass consent quiz)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
OUD treatment entry (number [%] of participants who enter OUD treatment) | 1 month
  The primary outcome for the trial is OUD treatment entry by 1 month post-enrollment, defined as admission to a buprenorphine provider (either office-based care or a specialty OUD program), or other licensed OUD treatment program (e.g., methadone, medical detox followed by behavioral treatment).

SECONDARY OUTCOMES:
OUD treatment retention | 6 months
  Treatment retention will be examined as a secondary outcome and will be determined by self-report, with confirmation of admission/discharge dates through provider records if available.
Opioid use (self-report) | 6 months
  Self-reported days of opioid use in the past 30 days
Opioid use (urine test) | 6 months
  Opioid urine drug test
Cocaine use (self-report) | 6 months
  Self-reported days of cocaine use in the past 30 days
Cocaine use (urine test) | 6 months
  Cocaine urine drug test
OUD diagnostic criteria | 6 months
  Opioid use disorder diagnostic criteria will be assessed using items from the OUD criteria checklist derived from the modified World Mental Health-Composite International Diagnostic Interview (WMH-CIDI) items that map to the diagnostic criteria. The time frame of the criteria will be modified to past 30 days to capture acute changes.
Opioid overdose | 6 months
  Participants will be asked at follow-up about non-fatal opioid overdose experiences. We will obtain medical examiner reports to confirm fatal overdoses.
New Diagnoses of HIV/STIs | 6 months
  New diagnoses of HIV and sexually transmitted infections will be determined via self-report and health department records.
Adherence to recommended HIV/STI treatment | 6 months
  Participants will be asked at follow-up whether they took as directed their specific HIV/STI medications, including (if applicable) any extended antibiotics for bacterial STDs, antiretroviral therapy for HIV+ participants, and PrEP to safeguard against acquiring HIV.
Sex Risk Behaviors | 6 months
  Risky sex behaviors will be gauged by self-report, and include past 90 day frequency of unprotected sex and number of sex partners.
Drug Risk Behaviors | 6 months
  Risky drug injection practices in the past 90-days, gauged by self-report

CONTACTS AND LOCATIONS:
Overall Officials: Jan Gryczynski, Principal Investigator — Friends Research Institute, Inc.
Locations (2):
- United States (2):
  - Friends Research Institute, Baltimore, Maryland
  - Baltimore City Health Department Sexual Health Clinics, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified IPD and supporting documentation pending approval of an application and data use agreement with Friends Research Institute
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Access to de-identified data may be requested after publication of the primary and secondary outcome findings (approximately one year after study completion).
Access Criteria: 1. Application to Friends Research Institute.
  2. Approval of the application and secondary analysis protocol by Friends Research Institute.
  3. Execution of a data use agreement between the requesting party and Friends Research Institute.
  4. IRB-approval of the proposed secondary research protocol.

REFERENCES:
- [Derived] Nordeck CD, Sharma A, Terplan M, Dusek K, Gilliams E, Gryczynski J. Opioid Use Disorder Treatment Linkage at Strategic Touchpoints Using Buprenorphine (OUTLAST-B): Rationale, Design, and Evolution of a Randomized Controlled Trial. J Psychiatr Brain Sci. 2023;8(6):e230010. doi: 10.20900/jpbs.20230010. Epub 2023 Dec 25. PMID 38456042